CLINICAL TRIAL: NCT07237035
Title: Reclaiming Independence: Importance of Activities of Daily Living and Rehabilitation Objectives in Spinal Cord Injury Patients in Türkiye
Brief Title: Reclaiming Independence: Daily Activities and Rehabilitation Goals in Spinal Cord Injury
Status: Completed | Type: Observational
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Mucahit Atasoy, MD, Asst Prof, Medipol University
Other Study IDs: MedipolIU
Record Dates: First submitted 2025-11-13; First posted 2025-11-19 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Spinal Cord Injuries (SCI)
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Spinal Cord Injury: This observational group consists of 56 adults (aged 18-60) with Spinal Cord Injury (SCI) (either traumatic or non-traumatic, paraplegia or tetraplegia) . Participants are recruited from the Biruni University Physical Medicine and Rehabilitation clinics .

SUMMARY:
The purpose of this cross-sectional, observational survey was to assess the importance individuals with Spinal Cord Injury (SCI) in Türkiye place on specific Activities of Daily Living (ADL) and their target levels of independence for these activities after rehabilitation. The primary question it aims to answer is:

What are the functional priorities of individuals with SCI (e.g., eating, bathing, walking, wheelchair use), and what are their personal goals for independence in these activities?

Participants will complete a two-part questionnaire (at Biruni University Hospital) regarding the importance of ADL and independence goals.

DETAILED DESCRIPTION:
This study is a cross-sectional, single-center, observational study designed to address a recognized gap in rehabilitation literature concerning person-centered care in Spinal Cord Injury (SCI) . While aligning treatment with patient-specific goals is critical for improving motivation and adherence, most research identifying patient functional priorities has been conducted in Western populations . This research specifically aims to investigate these priorities within the Turkish SCI population, for which currently no data is available, thereby providing a foundation for culturally-relevant and patient-specific rehabilitation planning . The study will be conducted at the Biruni University Hospital Physical Medicine and Rehabilitation inpatient and outpatient clinics .

Participants and Data Collection Participants will complete a custom-designed two-part survey. In addition to the survey responses, relevant clinical and demographic data will be collected.

Survey Instrument: Activities of Daily Living Importance (ADLI) Questionnaire The primary data collection tool is the custom-designed, two-part ADLI Questionnaire. The ADL items were selected based on their relevance to the rehabilitation framework for SCI patients, covering self-care, mobility, and essential functional tasks.

Part 1: Functional Importance Assessment: This section assesses the patient's perceived importance of 10 key ADLs. Participants rate the significance of each ADL using an 10-point Visual Analog Scale (VAS) ranging from 0 (Not important at all) to 10 (Extremely important). The ADLs assessed include Eating, Bathing, Clean Intermittent Catheterization (Bladder emptying), Dressing, Oral/Face Care (Grooming), Sitting, Walking, Wheelchair Use, Transferring, and Sexual Activity.

Part 2: Assessment of Independence Goals: The second part of the survey assessed the participants' targeted post-rehabilitation independence levels for the specified 10 ADLs. Participants selected one of four mutually exclusive categories that reflect standard rehabilitation outcomes:

* Complete Independence (can perform without help),
* Modified Independence (requires an assistive device),
* Assisted (requires personal assistance),
* Total Dependence (unable to perform the activity).

Statistical Analysis: The data were analyzed using the SPSS Statistics 22.0 program. The normality of continuous variables was assessed using the Shapiro-Wilk test. For variables showing a normal distribution, independent samples t-tests and one-way ANOVA were used for group comparisons. For data that did not show a normal distribution, the Mann-Whitney U and Kruskal-Wallis tests were applied. The chi-square test was used for the analysis of categorical data; the Fisher exact test was used when the test conditions could not be met. The statistical significance level was set at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 18-60
* Tetraplegic or paraplegic due to spinal cord injury
* At least 1 month has passed since the rehabilitation begining
* Patients who agree to participate in the study and provide written consent

Exclusion Criteria:

* Having a disability due to any previous neurological (stroke, MS, Parkinson's, etc.) or orthopedic (amputation, knee prosthesis, etc.) reasons
* Insufficient mental functions to answer all questions

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The source population for this observational, cross-sectional study is the adult patient population with Spinal Cord Injury (SCI), both traumatic and non-traumatic, receiving care at a single-center academic setting in Turkey. Specifically, participants will be recruited from the inpatient and outpatient clinics of the Physical Medicine and Rehabilitation Department at Biruni University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2025-11-03 (Actual); Primary Completion 2026-01-03 (Actual); Study Completion 2026-01-15 (Actual)

PRIMARY OUTCOMES:
Perceived Importance of Activities of Daily Living (ADLs) Assessed by Visual Analog Scale (VAS) | Baseline
  The primary outcome is the quantitative score representing the perceived importance of 10 specific Activities of Daily Living (ADLs) (e.g., Eating, Bathing, Transfer, Wheelchair Use) . Participants will rate each ADL using an 10-point Visual Analog Scale (VAS) , where 0 represents 'Not important at all' and 10 represents 'Extremely important' . The mean VAS score for each ADL will be calculated to identify the patient's functional priorities. This data will be collected via the custom-designed Activities of Daily Living Importance (ADLI) Questionnaire.

SECONDARY OUTCOMES:
Post-Rehabilitation İndependence Goals for ADLs | Baseline
  Assessment of the participant's stated personal rehabilitation goals for the same 10 ADLs. Goals are categorized using a 4-level nominal scale:
  Complete Independence (can perform without help), Modified Independence (requires an assistive device), Assisted (requires personal assistance), Total Dependence (unable to perform the activity).

CONTACTS AND LOCATIONS:
Overall Officials: Evrim Coşkun, MD Prof, Study Chair — Başakşehir Çam & Sakura City Hospital
Locations (1):
- Biruni University Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD), including all demographic, clinical, and primary/secondary outcome measures (VAS scores for ADL importance and targeted independence levels), will be shared with qualified researchers. The sharing period will commence 9 months after article publication and conclude 3 years thereafter. Data access requests must be accompanied by a methodologically sound proposal and will be granted upon the corresponding author's approval and the execution of a Data Use Agreement (DUA) to strictly ensure confidentiality and adherence to ethical guidelines.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 3 years following article publication.
Access Criteria: Qualified researchers who submit a methodologically sound proposal for achieving the goals of the approved proposal.

REFERENCES:
- [Background] Agarwal P, Mishra AN, Sudesh W, Prachir M, Dhananjaya S. Priorities of desired functional recovery in Indian spinal cord injury patients. J Clin Orthop Trauma. 2020 Sep-Oct;11(5):896-899. doi: 10.1016/j.jcot.2019.08.001. Epub 2019 Aug 1. PMID 32879577
- [Background] Ullah S, Qureshi AZ, AlWehaibi TA, Rathore FA, Sami W, Ayaz SB, AlKeid NH, Alibrahim MS, AlHabter AM, Alketheeri WB, Bashir MS. Functional priorities of individuals with spinal cord injury: a Saudi Arabian perspective. Spinal Cord. 2024 Sep;62(9):539-545. doi: 10.1038/s41393-024-01018-0. Epub 2024 Jul 26. PMID 39060481
- [Background] Ditunno PL, Patrick M, Stineman M, Ditunno JF. Who wants to walk? Preferences for recovery after SCI: a longitudinal and cross-sectional study. Spinal Cord. 2008 Jul;46(7):500-6. doi: 10.1038/sj.sc.3102172. Epub 2008 Jan 22. PMID 18209742